CLINICAL TRIAL: NCT00739765
Title: Psychotherapies for Chronic Post-Traumatic Stress Disorder
Brief Title: Effectiveness of Three Different Psychotherapies for Chronic Post-Traumatic Stress Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, John Markowitz, Clinical Psychiatrist, New York State Psychiatric Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: #5660, R01 MH079078; R01MH079078 (NIH)
Record Dates: First submitted 2008-08-20; First posted 2008-08-22 (Estimated); Results first posted 2015-11-16 (Estimated); Last update posted 2019-03-05 (Actual); Status verified 2019-02

CONDITIONS: Post-Traumatic Stress Disorder
Keywords: Trauma; Psychotherapy; Anxiety
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Wounds and Injuries; Anxiety Disorders | interventions — Interpersonal Psychotherapy; Relaxation Therapy

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial of three time-limited (14 week) psychotherapies for unmedicated patients with chronic posttraumatic stress disorder (PTSD)
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 Interpersonal Psychotherapy (IPT) (Experimental): Participants will receive interpersonal psychotherapy.
  Interventions: Behavioral: Interpersonal Psychotherapy
- 2 Prolonged Exposure (PE) (Active Comparator): Participants will receive prolonged exposure therapy.
  Interventions: Behavioral: Prolonged Exposure Therapy
- 3 Relaxation therapy (Active Comparator): Participants will receive relaxation therapy.
  Interventions: Behavioral: Relaxation Therapy

INTERVENTIONS:
Behavioral: Interpersonal Psychotherapy — 14 weekly 50-minute sessions of interpersonal psychotherapy, a time-limited treatment that focuses on interpersonal functioning and social supports
  Arms: 1 Interpersonal Psychotherapy (IPT)
Behavioral: Prolonged Exposure Therapy — Ten 90-minute sessions, distributed over 14 weeks, of prolonged exposure, which involves the repeated, detailed recounting of the trauma to develop a coherent narrative and repeated exposure to reminders of the trauma
  Arms: 2 Prolonged Exposure (PE)
Behavioral: Relaxation Therapy — Nine 90-minute sessions and one 30-minute session, distributed over 14 weeks, that focus on muscle relaxation to address the physical symptoms of PTSD
  Arms: 3 Relaxation therapy

SUMMARY:
This study will examine whether interpersonal psychotherapy is as effective in treating post-traumatic stress disorder as the established therapies of prolonged exposure and relaxation.

DETAILED DESCRIPTION:
Post-traumatic stress disorder (PTSD) is caused by a traumatic experience often involving physical harm or the threat of harm or death. The emotional numbness and traumatic flashbacks symptomatic of PTSD interfere with everyday life for approximately 7.7 million adults. Besides prescription drug treatment, only exposure-based therapies, like prolonged exposure (PE) therapy, have been proved effective in treating PTSD. Interpersonal psychotherapy (IPT), which is not based on exposure, is effective in treating mood disorders, and pilot studies indicate it may also be effective in treating PTSD. IPT treats patients by helping them to improve their interpersonal functioning, as opposed to PE, which helps patients by guiding them to recreate traumatic memories in safe circumstances. This study will determine whether IPT is as effective as PE, the gold standard, in treating PTSD. Relaxation therapy, a commonly used control therapy for studies of PTSD, will be used for that purpose here.

All participants will be screened for PTSD, with those meeting the criteria being randomly assigned to one of the following three treatment groups:

* Group 1 participants will receive IPT. They will meet weekly for fourteen 50-minute sessions focusing on interpersonal consequences of the trauma affecting them and their relationships with others.
* Group 2 participants will receive PE. They will meet for 10, unevenly spaced 90-minute sessions during which they will face the trauma responsible for their symptoms.
* Group 3 participants will receive relaxation therapy. They will meet for nine 90-minute sessions and one 30-minute session during which they will learn relaxation methods.

All treatments will last 14 weeks, with assessments made by mental health professionals at screening, the midpoint of the study, the end of the study, and a 3-month follow-up. PTSD symptoms will be assessed through clinical interviews and self-report measures. In addition, participants will complete other interviews and tests that will examine a variety of factors relating to mental health, including comorbidity of other conditions, affect, social functioning, and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Meets DSM-IV (Diagnostic and Statistical Manual of Mental Disorders) criteria for primary, chronic PTSD
* At least moderately severe symptoms, defined by a minimum total (frequency plus severity) Clinician-Administered PTSD Scale score greater than 50
* Willing to undergo an independent clinical assessment and other ratings

Exclusion Criteria:

* Diagnosis of schizophrenia, bipolar disorder, or other psychotic disorders
* Psychiatric disorder due to a general medical condition
* Current substance abuse or dependence
* Acute suicide or homicide risk
* Unstable or life-threatening medical condition
* Primary diagnosis of borderline personality disorder, major depressive disorder, or major depression, melancholic subtype
* Diagnosis of antisocial personality disorder
* At least partial benefit from current treatment regimen
* Unwillingness to discontinue current ineffective psycho- or pharmacotherapy
* Inability to speak or read English

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2008-04; Primary Completion 2013-03 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John C. Markowitz, MD, Principal Investigator — New York State Psychiatric Institution
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bleiberg KL, Markowitz JC. A pilot study of interpersonal psychotherapy for posttraumatic stress disorder. Am J Psychiatry. 2005 Jan;162(1):181-3. doi: 10.1176/appi.ajp.162.1.181. PMID 15625219
- [Background] Markowitz JC, Bleiberg KL, Christos P, Levitan E. Solving interpersonal problems correlates with symptom improvement in interpersonal psychotherapy: preliminary findings. J Nerv Ment Dis. 2006 Jan;194(1):15-20. doi: 10.1097/01.nmd.0000195314.80210.41. PMID 16462550
- [Background] Taylor S, Thordarson DS, Maxfield L, Fedoroff IC, Lovell K, Ogrodniczuk J. Comparative efficacy, speed, and adverse effects of three PTSD treatments: exposure therapy, EMDR, and relaxation training. J Consult Clin Psychol. 2003 Apr;71(2):330-8. doi: 10.1037/0022-006x.71.2.330. PMID 12699027
- [Background] Markowitz JC, Milrod B, Bleiberg K, Marshall RD. Interpersonal factors in understanding and treating posttraumatic stress disorder. J Psychiatr Pract. 2009 Mar;15(2):133-40. doi: 10.1097/01.pra.0000348366.34419.28. PMID 19339847
- [Background] Markowitz JC, Kaplowitz M, Suh EJ, Meehan KB, Neria Y, Jonker H, Rafaeli A, Lovell K. Treating patients who strain the research psychotherapy paradigm. J Nerv Ment Dis. 2012 Jul;200(7):594-7. doi: 10.1097/NMD.0b013e31825bfaf4. PMID 22759936
- [Background] Amsel LV, Hunter N, Kim S, Fodor KE, Markowitz JC. Does a study focused on trauma encourage patients with psychotic symptoms to seek treatment? Psychiatr Serv. 2012 Apr;63(4):386-9. doi: 10.1176/appi.ps.201100251. PMID 22476306
- [Background] Rafaeli AK, Markowitz JC. Interpersonal psychotherapy (IPT) for PTSD: a case study. Am J Psychother. 2011;65(3):205-23. doi: 10.1176/appi.psychotherapy.2011.65.3.205. PMID 22032045
- [Background] Markowitz JC, Milrod BL. The importance of responding to negative affect in psychotherapies. Am J Psychiatry. 2011 Feb;168(2):124-8. doi: 10.1176/appi.ajp.2010.10040636. No abstract available. PMID 21297048
- [Background] Markowitz JC. IPT and PTSD. Depress Anxiety. 2010 Oct;27(10):879-81. doi: 10.1002/da.20752. No abstract available. PMID 20886608
- [Background] Markowitz JC, Lipsitz J, Milrod BL. Critical review of outcome research on interpersonal psychotherapy for anxiety disorders. Depress Anxiety. 2014 Apr;31(4):316-25. doi: 10.1002/da.22238. Epub 2014 Feb 3. PMID 24493661
- [Result] Markowitz JC, Petkova E, Neria Y, Van Meter PE, Zhao Y, Hembree E, Lovell K, Biyanova T, Marshall RD. Is Exposure Necessary? A Randomized Clinical Trial of Interpersonal Psychotherapy for PTSD. Am J Psychiatry. 2015 May;172(5):430-40. doi: 10.1176/appi.ajp.2014.14070908. Epub 2015 Feb 13. PMID 25677355
- [Result] Markowitz JC, Meehan KB, Petkova E, Zhao Y, Van Meter PE, Neria Y, Pessin H, Nazia Y. Treatment preferences of psychotherapy patients with chronic PTSD. J Clin Psychiatry. 2016 Mar;77(3):363-70. doi: 10.4088/JCP.14m09640. PMID 26115532
- [Result] Markowitz JC, Petkova E, Biyanova T, Ding K, Suh EJ, Neria Y. EXPLORING PERSONALITY DIAGNOSIS STABILITY FOLLOWING ACUTE PSYCHOTHERAPY FOR CHRONIC POSTTRAUMATIC STRESS DISORDER. Depress Anxiety. 2015 Dec;32(12):919-26. doi: 10.1002/da.22436. Epub 2015 Oct 6. PMID 26439430
- [Result] Markowitz JC, Neria Y, Lovell K, Van Meter PE, Petkova E. History of sexual trauma moderates psychotherapy outcome for posttraumatic stress disorder. Depress Anxiety. 2017 Aug;34(8):692-700. doi: 10.1002/da.22619. Epub 2017 Apr 4. PMID 28376282
- [Result] Markowitz JC, Choo TH, Neria Y. Do Acute Benefits of Interpersonal Psychotherapy for Posttraumatic Stress Disorder Endure? Can J Psychiatry. 2018 Jan;63(1):37-43. doi: 10.1177/0706743717720690. Epub 2017 Jul 25. PMID 28743198
- [Result] Suarez-Jimenez B, Zhu X, Lazarov A, Mann JJ, Schneier F, Gerber A, Barber JP, Chambless DL, Neria Y, Milrod B, Markowitz JC. Anterior hippocampal volume predicts affect-focused psychotherapy outcome. Psychol Med. 2020 Feb;50(3):396-402. doi: 10.1017/S0033291719000187. Epub 2019 Feb 18. PMID 30773148
- See also: Click here for more information on trauma and PTSD at the Web site of Columbia University Medical Center, New York State Psychiatric Institute — http://www.columbiatrauma.org/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 1 Interpersonal Psychotherapy (IPT) | 2 Prolonged Exposure (PE) | 3 Relaxation Therapy
Started | 40 | 38 | 32
Completed | 34 | 27 | 21
Not Completed | 6 | 11 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 1 Interpersonal Psychotherapy (IPT) | 2 Prolonged Exposure (PE) | 3 Relaxation Therapy | Total
Number analyzed (Participants) | 40 | 38 | 32 | 110
Age, Continuous [Mean (Standard Deviation); unit: Years] | 38.12 (11.21) | 41.76 (11.99) | 40.62 (11.48) | 40.10 (11.57)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 21 | 28 | 77
  Male | 12 | 17 | 4 | 33
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 12 | 11 | 31
  Not Hispanic or Latino | 32 | 26 | 21 | 79
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 3 | 2 | 4 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 4 | 9 | 6 | 19
  White | 31 | 22 | 19 | 72
  More than one race | 2 | 5 | 3 | 10
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 40 | 38 | 32 | 110

OUTCOME MEASURES:

1. Primary Outcome: Clinician-Administered PTSD Scale (CAPS)
Description: Continuous measure scale of PTSD symptoms severity. Generally considered state of the art. Range 0-136 (17 items each rated for frequency and for intensity, each on a 0-4 scale). Scores >50 indicate at least moderately severe PTSD; scores <20 were defined as remission. See Blake DD, Weathers FW, Nagy LM, et al: The development of a clinician-administered PTSD scale. J Trauma Stress 1995; 8:75-90; Weathers FW, Keane TM, Davidson JRT: Clinician-Administered PTSD Scale: a review of the first ten years of research. Depression and Anxiety 2001;13:132-156
Time Frame: After 14 weeks of treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 1 Interpersonal Psychotherapy (IPT) | 2 Prolonged Exposure (PE) | 3 Relaxation Therapy
Number analyzed (Participants) | 40 | 38 | 32
units on a scale
  Baseline | 68.9 (16.2) | 72.1 (18.2) | 68.9 (16.4)
  Week 14 | 39.8 (24.3) | 37.5 (28.8) | 46.5 (31.0)

2. Secondary Outcome: Hamilton Depression Rating Scale
Description: Continuous scale to measure depressive symptom severity with a potential range from 0 to 74. Higher scores indicate more severe depressive symptoms. Scores <8 are generally considered not depressed; 8-12 mildly depressed; 13-19 moderately depressed; 20 and greater, severely depressed. Reference: Hamilton M: A rating scale for depression. J Neurol Neurosurg Psychiatry 1960;25:56-62
Time Frame: After 14 weeks of treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 1 Interpersonal Psychotherapy (IPT) | 2 Prolonged Exposure (PE) | 3 Relaxation Therapy
Number analyzed (Participants) | 40 | 38 | 32
units on a scale
  Baseline | 18.3 (6.5) | 20.2 (6.7) | 21.0 (7.1)
  Week 14 | 13.8 (8.8) | 12.3 (8.8) | 14.8 (9.1)

ADVERSE EVENTS:
Time Frame: 14 weeks; treatment responders followed to 26 weeks.
Arm/Group | 1 Interpersonal Psychotherapy (IPT) | 2 Prolonged Exposure (PE) | 3 Relaxation Therapy
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/38 | 0/32
Other Adverse Events (participants affected / at risk) | 0/40 | 0/38 | 0/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1 Interpersonal Psychotherapy (IPT) (N=40) | 2 Prolonged Exposure (PE) (N=38) | 3 Relaxation Therapy (N=32)
Clinical deterioration/protocol violation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Limited generalizability of unmedicated sample; incomplete therapist fidelity rating; limited sample size.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes